CLINICAL TRIAL: NCT03938688
Title: Two-armed Single Blinded Non-inferiority Registry Based Randomized Control Trial Comparing Transfascial Sutures for Mesh Fixation to No Mesh Fixation for Open Retromuscular Repairs
Brief Title: Randomized Control Trial Comparing Transfascial Suture for Mesh Fixation to No Mesh Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ajita Prabhu, MD, Assistant Professor of Surgery, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-333
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ventral Hernia; Incisional Hernia
Keywords: ventral hernia repair; mesh; pain; incisional hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transfascial sutures for mesh fixation (Other): Mesh will be placed in the retromuscular space, with wide overlap on all sides. Full thickness transfascial sutures will be placed circumferentially to secure the mesh using slowly absorbable no. 1 sutures. A total of at least six transfascial sutures will be placed universally for all patients with additional sutures allowed according to each surgeon's discretion. Additional bone or ligament sutures for mesh fixation will be allowed according to each surgeon's discretion.
  Interventions: Procedure: Mesh placement with Transfascial Sutures
- No mesh fixation (No Intervention): Mesh will be placed in the retromuscular space, with wide overlap on all sides. No fixation method will be used. Bone or ligament sutures for mesh fixation will not be allowed.

INTERVENTIONS:
Procedure: Mesh placement with Transfascial Sutures — Sutures that pass through the full thickness of the abdominal wall, which are used routinely for mesh fixation
  Arms: Transfascial sutures for mesh fixation

SUMMARY:
This will be a single blinded, registry based, non-inferiority, randomized control trial comparing transfacial sutures for mesh fixation to no mesh fixation in open retromuscular repairs. The primary outcome of interest is recurrence measured one year postoperatively as per standard of care at Cleveland Clinic Center for Abdominal Core Health. Hence, recurrence will be measured using either physical examination, CT scan, or the Ventral Hernia Recurrence Inventory (VHRI). Study population will include all adult patients (18 years or older) undergoing elective open ventral hernia repair of a clean (Wound class I) defect, where the midline fascia can be approximated and mesh will be placed in the retromuscular position. Only a midline approach to hernia repair and hernia widths equal to or less than 20cm measured intraoperatively will be included

DETAILED DESCRIPTION:
The techniques of mesh fixation in open incisional hernia repair is an active area of discussion and debate. When first described, the posterior component separation with the transversus abdominis muscle release involved placing the mesh in the retromuscular space, and fixating it circumferentially with transfascial sutures. These sutures penetrate the entire length of the abdominal wall and can be a significant source of pain. This study aims to evaluate the effect of using no fixation on recurrence rates, compared to the standard of care of using transfacial sutures. The investigators hypothesize that recurrences rates for patients who receive no fixation will be non-inferior to those receiving transfascial sutures.

This will be a single blinded, registry based, non-inferiority, randomized control trial comparing transfacial sutures for mesh fixation to no mesh fixation in open retromuscular repairs. This will be a two-arm trial with intervention 1: intervention 2 and control allocation ratio of 1:1. The Americas Hernia Society Quality Collaborative (AHSQC) will serve as the platform for data collection. The AHSQC is a multicenter, nationwide quality improvement effort with the mission of improving the quality of hernia care. Data points not recorded in the AHSQC will be collected by a trained research coordination or research fellow and uploaded into a Research Electronic Data Capture (RedCAP®) database hosted at the Cleveland Clinic

Study population will include all adult patients (≥ 18 years) undergoing elective open ventral hernia repair, where the midline fascia can be approximated and mesh will be placed in the retromuscular position. Only a midline approach to hernia repair and hernia widths equal to or less than 20cm measured intraoperatively will be included. Exclusion criteria include patients unable to give consent, vulnerable populations, parastomal hernias, hernia width measuring more than 20cm intraoperatively, patients planned for minimally invasive approaches or open repairs with mesh placed in a position other than retromuscular, or those who were not able to undergo successful retromuscular mesh placement. Finally, open repairs performed through a different incision than the standard midline approach will also be considered exclusion criteria, as well as the inability to close the midline fascia.

Study Interventions:

* Intervention 1 (Control): Mesh will be placed in the retromuscular space, with wide overlap on all sides. Full thickness transfascial sutures will be placed circumferentially to secure the mesh using slowly absorbable no. 1 sutures. A total of six transfascial sutures will be placed universally for all patients with additional sutures allowed according to each surgeon's discretion. Additional bone or ligament sutures for mesh fixation will be allowed according to each surgeon's discretion.
* Intervention 2: Mesh will be placed in the retromuscular space, with wide overlap on all sides. No fixation method will be used. Bone or ligament sutures for mesh fixation will not be allowed.

Specific Aims:

* Aim 1: To investigate the non-inferiority of recurrence rates in patients receiving no fixation for a mesh placed in retromuscular position compared to those receiving circumferential transfascial suture fixation. Either physical examination, CT scan, or the Ventral Hernia Recurrence Inventory (VHRI) will be used to measure recurrence at one-year follow up.
* Aim 2: To determine if no mesh fixation results in less pain in the immediate postoperative period, measured by the Numeric Pain Rating Scale (NRS-11).
* Aim 3: To determine if no mesh fixation results in less pain on 30 day follow up, measured by using the Patient Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey
* Aim 4: To determine if in-hospital intravenous and oral opioid consumption will differ between those who received transfascial sutures and those who did not receive any fixation.
* Aim 5: To determine if length of stay will differ between those who received transfascial sutures and those who did not receive any fixation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective open ventral hernia repair, where the midline fascia can be approximated and mesh will be placed in the retromuscular position
* A midline approach to hernia repair
* Hernia widths equal to or less than 20cm measured intraoperatively

Exclusion Criteria:

* Patients unable to give consent and vulnerable populations.
* Parastomal hernias
* Hernia width measuring more than 20cm intraoperatively
* Patients planned for minimally invasive approaches or open repairs with mesh placed in a position other than retromuscular, or those who were not able to undergo successful retromuscular mesh placement.
* Open repairs performed through a different incision than the standard midline approach
* Inability to close the midline fascia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Recurrence | One year
  primary outcome of interest is recurrence measured one year postoperatively as per standard of care at the Cleveland Clinic Center for Abdominal Core Health. Hence, recurrence will be measured using either physical examination, CT scan, or the Ventral Hernia Recurrence Inventory (VHRI), either during a physical or a virtual clinic visit and/or using the telephone. The VHRI is a validated patient reported outcomes tool, a three-question survey that can be administered directly to patients without clinical interaction.

SECONDARY OUTCOMES:
Post-operative pain | Baseline and 30 day follow up. The 30-day follow up period will extend from 15 - 45 days postoperatively.
  Pain scores will be measured by Patient Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey. The PROMIS pain intensity 3a survery is a National Institute of Health-developed validated tool, which focuses on PROs of pain characteristics.
Post-operative pain | Baseline, first 7 days post-operatively, and 30 day follow up. The 30-day follow up period will extend from 15 - 45 days postoperatively.
  Pain scores will be measured using the Numeric Pain Rating Scale (NRS-11). The NRS-11 is Likert scale where the patient mark their current pain on scale from 1 to 10.
Daily opioid requirements | first 7 days of the post-operative period
  Opioid requirements will be assessed by measuring the cumulative dose of opioids administered intravenously (infused through a patient-controlled analgesia device as well as the quantity of opioids administered intravenously as rescue, if needed) and the quantity of opioids administered through oral preparations. The total dose of opioid consumption will be converted to morphine equivalence.
Length of stay | From date of admission to hospital until the date of discharge from hospital, assessed up to 60 weeks
  Length of in-hospital stay will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ajita S Prabhu, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Abdominal Core Health, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, rather the results of the aggregate groups of patients will be shared

REFERENCES:
- [Derived] Ellis RC, Petro CC, Krpata DM, Beffa LRA, Miller BT, Montelione KC, Maskal SM, Tu C, Huang LC, Lau B, Fafaj A, Rosenblatt S, Rosen MJ, Prabhu AS. Transfascial Fixation vs No Fixation for Open Retromuscular Ventral Hernia Repairs: A Randomized Clinical Trial. JAMA Surg. 2023 Aug 1;158(8):789-795. doi: 10.1001/jamasurg.2023.1786. PMID 37342018